CLINICAL TRIAL: NCT04677842
Title: European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC): Paediatric Protocol
Brief Title: European Pregnancy and Paediatric Infections Cohort Collaboration: Paediatric Protocol
Acronym: EPPICC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PENTA Foundation (Network)
Collaborators: University College, London (Other); Centre Hospitalier Universitaire Saint Pierre (Other); German Pediatric and Adolescent HIV Cohort (GEPIC), GERMANY (Unknown); Greece Cohort, GREECE (Unknown); Register for HIV infection in children, ITALY (Unknown); ATHENA ,THE NETHERLANDS (Unknown); Polish Paediatric Cohort, POLAND (Unknown); HSM/CHLN Lisbon, PORTUGAL (Unknown); Centro Hospitalar do Porto (Other); Victor Babes Hospital Cohort, Bucharest, ROMANIA (Unknown); Republican Hospital of Infectious Diseases, St Petersburg, RUSSIA (Unknown); Irkutsk AIDS Centre, RUSSIA (Unknown); The City HIV Centre, St Petersburg, RUSSIA (Unknown); CoRISpe-cat cohort of HIV-infected children, SPAIN (Unknown); CoRISpe-S cohort of HIV-infected children, SPAIN (Unknown); Karolinska Institutet (Other); Swiss Mother and Child HIV Cohort Study, SWITZERLAND (Unknown); Programs for HIV Prevention and Treatment (PHPT), THAILAND (Unknown); National Surveilliance of HIV in Pregnancy and Childhood and Collaborative HIV Paediatric Study (CHIPS) (Unknown); Collaborative HIV Paediatric Study (CHIPS) (Unknown); Ukraine Paediatric HIV Cohort, UKRAINE (Unknown)
Responsible Party: Sponsor
Other Study IDs: EPPICC
Record Dates: First submitted 2020-11-11; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: HIV Infections; Tuberculosis Infection; Hepatitis C; Covid19
Keywords: HIV; Tuberculosis; hepatitis C; COVID-19; paediatric; cohort; infectious diseases
MeSH Terms: conditions — HIV Infections; Latent Tuberculosis; Hepatitis C; COVID-19; Tuberculosis; Communicable Diseases | interventions — Art Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: ART Therapy
  Other Names: This is an observational study

SUMMARY:
Across Europe and worldwide, there are many studies following groups (cohorts) of children living with human immunodeficiency virus (HIV) and other infections over time, to monitor their long-term health. Some of these infections are rare: for example, few children in Western Europe are living with HIV, so the studies often have fairly small numbers of participants. This can make it difficult to answer research questions in these cohorts and means that doctors and researchers working with these patients in different countries need to work together. This is particularly important as children are not often included in clinical trials of treatments and other interventions.

The European Pregnancy and Paediatric Infections Cohort Collaboration (EPPICC) is an international network of researchers working together in this way. Researchers in the network represent cohort studies of pregnant women and children with, or at risk of, infections from across Europe and Thailand. The research focuses on infections in pregnant women and children, particularly HIV, hepatitis B and C virus, and tuberculosis, and, from 2020, novel coronavirus (COVID-19). By combining data from many cohorts, the researchers aim to answer questions that could not be answered by one study individually (for example, because a large number of pregnant women or children are needed to answer the question).

This protocol focuses on the paediatric component of EPPICC's research, which focuses on the treatment of children at risk of and living with infections. For example, what medicines are used most often and how do they affect children's health? EPPICC is an observational study, which means that children do not receive any extra treatment as part of the study. Instead, children are "observed" during their routine medical care. Each cohort keeps records of the children's health collected at routine clinic visits, including information such as date of birth and sex, results of diagnostic tests, treatments received, and any illnesses or other events that the children have had. The EPPICC study combines and analyses data from all of the cohorts that take part, to answer questions about the risks and benefits of different diagnosis or treatment strategies, the long-term effects of infection and treatment during childhood and young adulthood, and regional variations (e.g. between Western and Eastern Europe) in the risk and management of infections.

All of the data collected through the EPPICC Paediatric Protocol are stored securely at the Medical Research Council Clinical Trials Unit (MRC CTU) at UCL. Data collection and storage are governed by the General Data Protection Regulation. A Steering Committee guides the research to make sure it is relevant and of high quality. Public and patient involvement (PPI) may be provided by individual cohorts' own groups, as well as by the interlinked Penta organisation, which is a network of paediatricians and researchers working in infections in Europe and globally. The PPI groups help with release of the results of the research. The results are also published on the Penta Foundation's public website (https://penta-id.org/), and presented at conferences and published in Open Access scientific journals.

DETAILED DESCRIPTION:
MAIN AIM OF THE STUDY The overall aim of the EPPICC Paediatric Protocol is to analyse individual patient data from across collaborating European and international cohorts on infections in children and young people, to inform optimal prevention and treatment strategies.

MAIN AREAS OF FOCUS HIV: prevalence and incidence of immunological and virological failure, HIV resistance, AIDS and non-AIDS events, mortality, cascade of care, engagement in care (including after transfer to adult care); antiretroviral therapy status and toxicities (adverse events, serious adverse events and discontinuation of drug) HCV: disease progression, uptake and outcome (effectiveness and safety) of HCV treatment in HCV mono- and HCV-HIV co-infected patients TB: incidence (including exploration of different diagnostic/screening strategies across regions) of LTBI and TB disease; outcomes of TB treatment including treatment of LTBI COVID-19: prevalence and incidence of infection and disease among both the general population and specifically among children and adolescents living with HIV; admission to hospital/ICU; outcomes (including resolution, death, sequelae (e.g. paediatric inflammatory syndrome temporally associated with SARS-CoV-2)) COHORT / INVESTIGATOR INCLUSION CRITERIA The study Sponsor has overall responsibility for site and investigator selection.

The Principal Investigators of cohorts which have participated in previous EPPICC data mergers will be approached to ascertain their interest in participating in future data mergers. New cohorts may also be identified and may be invited to participate. The key inclusion criterion for a cohort to participate is enrolment of children and adolescents with the infection of interest. All cohorts who are able to commit to submitting and cleaning data, obtaining any ethical, regulatory or other approvals required locally, and completion of data sharing agreements in accordance with the project timelines will be included.

DATA COLLECTION Collected data are pseudonymised: no names, initials, hospital numbers, national ID or addresses of patients are collected. Core data items included in most EPPICC paediatric data mergers include the following; Demographic: Date of birth, sex, ethnicity/country of origin, country of residence Therapeutic: Prophylaxis and treatment data (HIV, HCV, TB and COVID-19 treatments) including start and stop dates, drug names, doses and frequency of administration, and reasons for change/discontinuation Diagnostic: Diagnostic tests for infections undertaken, including dates and results Concurrent treatments: Other medications Clinical Infection status: (HIV, TB, HCV, HBV, SARS-CoV-2, other infection of interest), mode of acquisition of infection, date of diagnosis, disease stage Clinical (other events): Adverse events (e.g. severity, causal relation to drugs), AIDS- and non-AIDS- defining malignancies, COVID-19 sequelae, weight, height, death, causes of death, pregnancy, hospitalisations Laboratory: Absolute CD4 counts and percentage, HIV RNA, HCV RNA measurements, other lab markers Other Follow-up status, reason for study drop-out, transfer to adult care

For certain analyses, additional data items may be requested, and may include:

* Biochemistry results
* Further details of severe adverse events
* Outcome of severe events. Data merger methods Individual cohorts collect data from medical records in clinics. Cohorts then send electronic datasets to the EPPICC Paediatric Data Manager, using a format and method defined in an EPPICC Standard Operating Procedure. For the ongoing HIV analyses, data variables are based on HICDEP data formats. HICDEP is the HIV Cohorts Data Exchange Protocol (www.hicdep.org) and is based on a relational structure, with data presented in a series of tables, together with the lookup tables for the codes to be used. For other future cohort collaborations, the variables to be collected and the database format will be based on existing data collection tools and standards where possible. Transfer of data to the EPPICC Paediatric Data Manager takes place using Galaxkey or an equivalent secured method.

Submitted data are subjected to a range of logic and consistency checks. STATISTICAL CONSIDERATIONS EPPICC analyses may cover a wide range of questions, although individual Concept Sheets are specific to focussed research questions.

SAMPLE SIZE Data are collected on all eligible participants enrolled in the participating centres who meet the inclusion criteria. Sample size calculations are carried out for specific planned analyses to ensure that sufficient participants are available to meaningfully answer each research question.

ANALYSIS PLAN Each Concept Sheet includes a brief analysis plan. Standard statistical methods are used in the analysis of different types of exposure and outcome data. Adjustment for confounding may be achieved through multivariable modelling or using alternative approaches such as propensity scoring. Missing data are to be expected and, depending on the analysis and the amount and likely mechanisms of missing data, may be approached using complete case analysis or techniques such as multiple imputation. Details of specific analytical approaches are included in each Concept Sheet. Previous analyses of EPPICC paediatric data have used approaches including Cox regression, linear regression, logistic regression, and propensity score matching. Cohorts may be grouped by region (as cohorts within the same region are often similar in terms of epidemiology and treatment approaches), and region is then included as a covariate in the analysis.

REGULATORY & ETHICAL ISSUES COMPLIANCE EPPICC is an observational study with no study-specific interventions beyond those received in routine care. Nevertheless, it is conducted in compliance with the approved protocol, the Declaration of Helsinki 1996, the principles of Good Clinical Practice, the General Data Protection Regulation and the UK Data Protection Act 2018 (DPA number: Z6364106), and the UK Policy Framework for Health and Social Care Research.

Each cohort is responsible for ensuring compliance with local and national regulatory and ethical processes.

DATA RETENTION

The paediatric study dataset will be stored at the MRC CTU at UCL, in accordance with national data legislation. A final copy will be sent to the study sponsor, the Penta Foundation. The dataset will be held for a minimum of 5 years after the end of the study.

DATA SHARING AGREEMENTS BETWEEN COHORTS AND EPPICC Individual cohorts, the Penta Foundation and the MRC CTU at UCL are required to sign a Data Sharing Agreement (DSA), which allows transfer of data between cohorts and the Penta Foundation and the MRC CTU at UCL. All data will be handled and used in accordance with the DSA. Cohorts should return the DSA, once signed, to the project coordinator at the Penta Foundation.

THIRD PARTY DATA SHARING REQUESTS Extracts of EPPICC data may be requested for other cohort collaboration analyses, both nationally and internationally. Requests to access EPPICC data will be considered on a case by case basis. Transfer of EPPICC data (partial or complete) to third party collaborators requires approval from the PIs of cohorts contributing data (or authorised cohort representatives) and is subject to a contract and Data Sharing Agreement, if applicable. All data transfer is conducted through a secure process. Any data transferred to third parties must be stored by third parties in compliance with all relevant data protection regulations.

Researchers wishing to access EPPICC data should contact the EPPICC Study Team in the first instance. A Concept Sheet is then required, which would be circulated to and discussed with all potential contributing cohorts.

ELIGIBILITY:
Children and adolescents diagnosed with HIV and/or chronic HCV are eligible for inclusion in this data merger provided they meet one, or both, of the inclusion criteria below:

Children and young people living with HIV:

* Diagnosis of HIV infection at age <18 years
* ≥1 visit in paediatric care AND / OR
* Children and young people living with HCV:
* Diagnosis of chronic HCV infection at age <18 (defined as ≥1 antibody HCV positive results at ≥18 months of age or ≥1 HCV RNA positive result at ≥6 months of age) ≥1 visit in paediatric care

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Paediatric infectious disease clinics across Europe and Thailand
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
CD4 count in adulthood of young people with HIV assessed using routine clinical data | through study completion, an average of 5 year
2. Viral suppression in adulthood of young people with HIV assessed using routine clinical data | through study completion, an average of 5 year
Viral suppression defined as <50 copies, <400 copies and 1000 copies/mL) upto 144 weeks. | up to 144 weeks
CD4 change from drug start up to 144 weeks | up to 144 weeks
Cumulative incidence of virological failure (>1000 copies/mL) | through study completion, an average of 5 years
From start of novel drug of interest through to earliest date of the following: death, loss to follow-up, discontinuation of drug or last visit | From date of novel drug initiation until earliest date of death, loss to follow-up, discontinuation of drug or last visit assessed up to 36 months

IPD SHARING:
Plan to Share IPD: No